CLINICAL TRIAL: NCT01674478
Title: Early Supplementation of Enteral Microlipid With and Without Fish Oil in Premature Infants With Enterostomies
Acronym: EMLFO-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00021481
Record Dates: First submitted 2012-08-18; First posted 2012-08-28 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Prematurity; Intestine Perforation; Necrotizing Enterocolitis (NEC); Short Bowel Syndrome (SBS)
Keywords: NEC, SBS, enterostomy, fish oil, Microlipid, Intralipid,; enteral fat
MeSH Terms: conditions — Premature Birth; Intestinal Perforation; Enterocolitis, Necrotizing; Short Bowel Syndrome | interventions — Safflower Oil; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Microlipid with fish oil group (Experimental): This group will be given early enteral lipid supplementation with Microlipid and fish oil.
  Interventions: Dietary Supplement: Microlipid with fish oil
- Microlipid group (Active Comparator): This group will be given early enteral lipid supplementation only with Microlipid.
  Interventions: Dietary Supplement: Microlipid

INTERVENTIONS:
Dietary Supplement: Microlipid with fish oil — Fish oil will start with initial feeding after ostomy placement and Microlipid will start once infant tolerating enteral feeds at 20 ml /kg/d while weaning the Intralipid, which both will be continued until reanastomosis.
  Arms: Microlipid with fish oil group
Dietary Supplement: Microlipid — A small amount (ml) of Microlipid to match the amount of fish oil in ML/FO group will start with initial feeding after ostomy placement and Microlipid will start once infant tolerating enteral feeds at 20 ml /kg/d while weaning the Intralipid, which will be continued until reanastomosis.
  Arms: Microlipid group

SUMMARY:
Necrotizing enterocolitis (NEC) and spontaneous intestinal perforation (SIP) are common devastating gastrointestinal diseases in premature infants. These infants often need surgical intervention to remove the dead bowel and create temporary enterostomies, resulting in short bowel syndrome (SBS), a malabsorption state due to insufficient bowel length or dysfunction to digest and absorb nutrients adequately.

These infants are often nourished primarily with parental nutrition (PN) which can lead to many complications including PN-associated liver disease. However, with enteral feeding, the remaining bowel can adapt somewhat to the shortened state, reducing the need for PN. Enteral fats appear to be the most trophic macronutrients with the long chain polyunsaturated fatty acids (LCPUFA) being the most beneficial in promoting bowel adaptation.

Fish oil (FO), a main source of n-3 LCPUFA, has been shown to promote bowel adaptation. Microlipid (ML) primarily contains n-6 PUFA and has been found to decrease ostomy output and increase weight gain in some SBS infants. WThe investigators will soon have completed a randomized clinical trial (EMLFO trial) (WFUHS IRB00011501, NCT01306838) entitled "Early Supplementation of Enteral Lipid with Combination of Microlipid and Fish Oil in Infants with Enterostomies". The preliminary data suggest that (a) by supplementing enteral ML/FO, we were able to decrease the use of IL; (b) premature infants in the treatment group who received ML/FO achieved higher enteral calorie (% of total calorie) intake before reanastomosis and better weight gain (g/day) after reanastomosis than those who received routine care in control group; and (c) the direct bilirubin level before reanastomosis tended to be lower in the treatment group than the control group although the difference was not statistically significant. Because the intervention consisted of both an increase in enteral fat intake as well as a specific type of fat intake (i.e. FO), it is unclear whether improved outcomes in the ML/FO group are attributable to FO's anti-inflammatory effects or the increased fat intake. Therefore, the investigators have designed a next randomized clinical trial to compare ML alone versus ML plus FO. We hypothesize that as compared to ML alone, ML plus FO will result in decreased systemic inflammation, as indicated by blood levels of inflammation-related proteins and indicators of oxidative stress.

DETAILED DESCRIPTION:
In comparison to EMLFO trial, the EMLFO-2 study will modify the eligibility criteria to only enroll the infants who have birthweight equal to or less than 1250 g with a jejunostomy or ileostomy as the result of surgical treatment for small intestine perforation or NEC in order to increase the homogeneity of patient population.

ELIGIBILITY:
Inclusion Criteria:

1. infants (age range: newborn to ≤ 2-month-old) whose birth weight are ≤ 1250g;
2. who are admitted to BCH NICU for surgical intervention for NEC or small intestine perforation and then to have a jejunostomy or ileostomy;
3. who are expected to need full or partial PN for at least 21days from the day of ostomy placement; and
4. who have received enteral feedings ≤ 4 days since ostomy placement.

Exclusion Criteria:

1. infant with birth weight > 1250g;
2. infant with colostomy;
3. infants with enterostomy but

   * unable to obtain written informed consent from parent;
   * presence of congenital liver, renal, or metabolic diseases or syndromes or perinatal asphyxia;
   * ostomy caused by surgical treatment for a condition other than NEC or small intestine perforation; and
   * unable to initiate enteral feeding for more than 28 days since ostomy placement.

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-03-17 (Actual); Study Completion 2015-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qing Yang, MD, PhD, Principal Investigator — WFUHS
Locations (1):
- Wake Forest University Health Science, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Yang Q, Kock ND. Effects of dietary fish oil on intestinal adaptation in 20-day-old weanling rats after massive ileocecal resection. Pediatr Res. 2010 Sep;68(3):183-7. doi: 10.1203/PDR.0b013e3181eb2ee5. PMID 20531250
- [Background] Yang Q, Lan T, Chen Y, Dawson PA. Dietary fish oil increases fat absorption and fecal bile acid content without altering bile acid synthesis in 20-d-old weanling rats following massive ileocecal resection. Pediatr Res. 2012 Jul;72(1):38-42. doi: 10.1038/pr.2012.41. Epub 2012 Mar 23. PMID 22447320
- [Result] Yang Q, Welch CD, Ayers K, Turner C, Pranikoff T. Early enteral fat supplementation with microlipid(R) and fish oil in the treatment of two premature infants with short bowel. Neonatology. 2010;98(4):348-53. doi: 10.1159/000316067. Epub 2010 Oct 27. PMID 20980771
- [Result] Woods CW, Ayers K, Turner C, Pranikoff T and Qing Yang. A Novel Nutritional Approach to Prevent Parenteral Nutrition-Associated Cholestasis in Two Premature Infants with Short Bowel Syndrome. ICAN: Infant, Child, & Adolescent Nutrition 2013 5: 32-36.
- [Result] Yang Q, Ayers K, Chen Y, Helderman J, Welch CD, O'Shea TM. Early enteral fat supplement and fish oil increases fat absorption in the premature infant with an enterostomy. J Pediatr. 2013 Aug;163(2):429-34. doi: 10.1016/j.jpeds.2013.01.056. Epub 2013 Feb 28. PMID 23453547

RESULTS

PARTICIPANT FLOW:
Groups:
- Microlipid and Fish Oil Group: This group will be given early enteral lipid supplementation with Microlipid and fish oil.
  Microlipid and fish oil: Fish oil will start with initial feeding after ostomy placement and Microlipid will start once infant tolerating enteral feeds at 20 ml /kg/d while weaning the Intralipid, which both will be continued until reanastomosis.
Period: Overall Study
Arm/Group | Microlipid and Fish Oil Group | Microlipid Group
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Microlipid and Fish Oil Group | Microlipid Group | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: weeks] — values represent the gestational age
  weeks | 26.3 (2.0) | 25.9 (2.0) | 26.1 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: The Serum Biomarkers of Inflammatory Cytokines
Description: Compare the serum biomarkers of inflammatory cytokines of the infants receiving ML/FO to the infants only receiving ML between the initial feeding after placement of an ostomy and reanastomosis
Time Frame: 2 years and 5 months
Population: No data collected
Arm/Group | Microlipid and Fish Oil Group | Microlipid Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Average Enteral Calorie (Total Calorie) Intake Before Reanast
Description: To compare the average enteral calorie (total calorie) intake of infants receiving ML/FO to the group only receiving ML between the initial feeding after placement of an ostomy and reanastomosis
Time Frame: 2 years and 5 months
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | Microlipid and Fish Oil Group | Microlipid Group
Number analyzed (Participants) | 9 | 9
kcal/kg/day | 52.1 (23.6) | 56.7 (15.6)

3. Secondary Outcome: The Average Weight Gain (g/Day) After Reanastomosis
Description: To compare the the average weight gain (g/day) of infants receiving ML/FO to the infants only receiving ML after reanastomosis
Time Frame: 2 years and 5 months
Measure: Mean (Standard Deviation); unit: g/d
Arm/Group | Microlipid and Fish Oil Group | Microlipid Group
Number analyzed (Participants) | 9 | 8
g/d | 26.6 (8.5) | 20.9 (12.2)

4. Primary Outcome: The Serum Biomarkers of Oxidative Stress
Description: Compare the serum biomarkers of oxidative stress of the infants receiving ML/FO to the infants only receiving ML between the initial feeding after placement of an ostomy and reanastomosis
Time Frame: 2 years and 5 months
Population: No data collected
Arm/Group | Microlipid and Fish Oil Group | Microlipid Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years and 5 months
Arm/Group | Microlipid and Fish Oil Group | Microlipid Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes